CLINICAL TRIAL: NCT04884308
Title: Effects of BCG Vaccine on the Immune System of Individuals With Cystic Fibrosis, Non-Cystic Fibrosis Bronchiectasis, and Healthy Volunteers
Brief Title: Bacille Calmette-Guerin (BCG) Vaccine for Immune Protection Against Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00256425
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis; Bronchiectasis Adult; Non-Tuberculous Mycobacteria
Keywords: BCG vaccine; Cystic fibrosis; Bronchiectasis; Non-tuberculosis mycobacteria
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cystic Fibrosis (Experimental): Participants with Cystic Fibrosis.
  Interventions: Biological: BCG TICE Vaccine
- Non Cystic Fibrosis Bronchiectasis (Experimental): Participants with Non Cystic Fibrosis Bronchiectasis.
  Interventions: Biological: BCG TICE Vaccine
- Healthy Volunteer (Active Comparator): Participants with no condition (healthy volunteers).
  Interventions: Biological: BCG TICE Vaccine

INTERVENTIONS:
Biological: BCG TICE Vaccine — Intradermal vaccination with BCG TICE

SUMMARY:
This is pilot study of the immunologic effects of intradermal Bacille Calmette-Guerin (BCG) vaccination of adults with cystic fibrosis (CF), non-CF bronchiectasis (NCFB), and healthy volunteers.

DETAILED DESCRIPTION:
This single-site, open-label clinical trial to investigate the immune effects of BCG vaccination in adults with cystic fibrosis, non-cystic fibrosis bronchiectasis and healthy volunteers by measuring pre and post vaccination immune responses, BCG uptake and protection against infections, including nontuberculous mycobacteria (NTM). This study will also gather data on study feasibility, tolerability, and safety.

ELIGIBILITY:
Inclusion Criteria (CF and non-CF bronchiectasis):

* Confirmed diagnosis of either CF or non-CF bronchiectasis
* Forced expiratory volume over one second (FEV1) > 40%
* Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained.
* Available for the study duration, including all planned follow-up visits

Inclusion Criteria (Healthy Volunteers):

* Negative HIV enzyme-linked immunosorbent assay (ELISA) and confirmatory test at screening.
* Willingness to participate in the study after all aspects of the protocol have been explained and written informed obtained.
* Available for the study duration, including all planned follow-up visits

Exclusion Criteria (All arms):

* Current or prior history of active or latent tuberculosis (TB) (per report, not formally tested) or NTM infection
* Prior BCG vaccination
* Previous vaccine in the past 4 weeks
* History of severe anaphylaxis to any vaccine or vaccine components
* History of organ/bone marrow transplantation or other immunosuppressing condition, including HIV
* Immunosuppressing drugs (including oral corticosteroids equivalent to >10mg of prednisone for 5 days) in the 30 days prior to study enrollment
* Cirrhosis or portal hypertension
* Pregnant or breastfeeding
* Receipt of another investigational product in the last 28 days or planned receipt during this study
* Has any other condition that, in the opinion of the principal investigator, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Lecthzin, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cystic Fibrosis | Non Cystic Fibrosis Bronchiectasis | Healthy Volunteer
Started | 14 | 2 | 14
Completed | 14 | 2 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data is presented for all patients enrolled that received BCG vaccination (N=30)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cystic Fibrosis | Non Cystic Fibrosis Bronchiectasis | Healthy Volunteer | Total
Number analyzed (Participants) | 14 | 2 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (13.5) | 44.4 (22.3) | 35.8 (10.2) | 34.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 6 | 13
  Male | 8 | 1 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 4
  White | 13 | 2 | 9 | 24
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 2 | 14 | 30
SFU count [Mean (Standard Deviation); unit: Spot forming units (SFU)] — Spot forming units (SFU) is a measure of immune response of mononuclear cells in response to M. avium lysate. Higher values indicate a stronger immune response.
  Spot forming units (SFU) | 35.22 (35.18) | 32.5 (17.68) | 38.75 (48.14) | 35.49 (33.67)

OUTCOME MEASURES:

1. Primary Outcome: BCG Uptake
Description: Change in concentration of interferon (IFN) gamma levels in blood after Bacille Calmette-Guérin (BCG) incubation relative to baseline as measured by SFUs. Spot forming units (SFU) is a measure of immune response of mononuclear cells in response to M. avium lysate. Higher values indicate a stronger immune response.
Time Frame: 3 months
Population: Analyzed all participants enrolled
Measure: Mean (Standard Error); unit: spot forming units
Arm/Group | Cystic Fibrosis | Non Cystic Fibrosis Bronchiectasis | Healthy Volunteer
Number analyzed (Participants) | 14 | 2 | 14
spot forming units | 48.06 (23.52) | 0.84 (16.92) | 35.97 (23.64)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cystic Fibrosis | Non Cystic Fibrosis Bronchiectasis | Healthy Volunteer
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/2 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/2 | 0/14
Other Adverse Events (participants affected / at risk) | 12/14 | 1/2 | 12/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cystic Fibrosis (N=14) | Non Cystic Fibrosis Bronchiectasis (N=2) | Healthy Volunteer (N=14)
Injection site pain (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 10 (10)
Swelling (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 2 (2)
pustule (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT04884308/Prot_SAP_000.pdf